CLINICAL TRIAL: NCT05166603
Title: Expanding Access to Comprehensive Geriatrics Care Via Telehealth (QUE 20-010)
Brief Title: Expanding Access to Comprehensive Geriatrics Care Via Telehealth
Acronym: TeleGRACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QUX 21-007; QUE HX0003205-01 (Other Grant/Funding Number: VA HSRD QUERI)
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Geriatric Syndrome
Keywords: comprehensive geriatrics assessment; telehealth; home visit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TeleGRACE (Experimental): Patients receive a virtual home visit and care from the GRACE team
  Interventions: Other: TeleGRACE
- Usual Care (No Intervention): Patients receive usual care

INTERVENTIONS:
Other: TeleGRACE — Patients receive a virtual home visit and care from the GRACE team
  Arms: TeleGRACE

SUMMARY:
The overall objective of the TeleGRACE project is to improve the care and outcomes of older Veterans with a recent inpatient stay by expanding access to the evidence-based GRACE program, by evaluating a telehealth implementation.

DETAILED DESCRIPTION:
The TeleGRACE evaluation will focus on three primary aims and a secondary aim:

Primary Aim 1: To examine the effectiveness of the TeleGRACE program, the investigators designed a randomized controlled implementation trial (RCT) powered for the primary outcome of 90-day all-cause mortality. The investigators will also examine its effectiveness for the secondary outcomes including 90-day readmissions, 1-year ED utilization (VA and non-VA), 1-year all-cause readmissions, 1-year mortality, as well as patient, caregiver, and staff satisfaction. The investigators hypothesize that patients who receive TeleGRACE will have lower 90-day mortality than patients in usual care.

Primary Aim 2: to examine the implementation of the TeleGRACE program. The implementation strategy is reflecting & evaluating. Implementation outcomes are based on the REAIM framework and include reach, efficacy (Aim 1), and implementation (total number of Veterans served, fidelity).

Primary Aim 3: to conduct a business-case analysis (BCA). The business case analysis will calculate the net financial savings or loss for TeleGRACE as the difference in the overall intervention costs and savings due to downstream benefits for patients receiving TeleGRACE versus usual care controls.

ELIGIBILITY:
Inclusion Criteria:

* Veterans discharged from the Indianapolis VA medical center (VAMC) for an medical/surgical diagnosis (excludes substance use disorder-related admissions; excludes planned admissions) within the prior week
* Age 70 years
* Not enrolled in home-based primary care (HBPC)
* Not enrolled in hospice
* Not in dialysis
* Primary care visit within VA in the prior 2 years
* Not residing in nursing home, skilled nursing facility, or CLC.
* Living >20 miles but <60 miles from the Indianapolis VAMC facility
* CAN score 95th percentile for mortality or missing CAN score
* Discharged from the hospital alive

Exclusion Criteria:

* Patients who have been randomized to the control arm after their index hospitalization who become readmitted to the hospital may not be re-randomized.
* By definition, GRACE patients are not eligible for TeleGRACE due to the drive distance >20 miles from the Indianapolis VAMC
* Enrolled in home-based primary care (HBPC)
* Enrolled in hospice
* Dialysis (hemodialysis or peritoneal dialysis)
* Residing in nursing home, skilled nursing facility, or CLC.
* Living <20 miles or 60 miles from the Indianapolis VAMC facility

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Bravata, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TeleGRACE | Usual Care
Started | 73 | 38
Completed | 5 | 38
Not Completed | 68 | 0
Not completed — Withdrawal by Subject | 68 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TeleGRACE | Usual Care | Total
Number analyzed (Participants) | 73 | 38 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 73 | 38 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.7 (6.1) | 77.0 (5.7) | 77.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 73 | 38 | 111
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 73 | 38 | 111

OUTCOME MEASURES:

1. Primary Outcome: 90-day All-cause Mortality
Description: The primary outcome is 90-day all-cause mortality measured from the date of discharge from the index hospitalization.
Time Frame: 90-days from discharge from the index hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | TeleGRACE | Usual Care
Number analyzed (Participants) | 5 | 38
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 90-days
Description: All unexpected, serious adverse events will be recorded
Arm/Group | TeleGRACE | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/38
Other Adverse Events (participants affected / at risk) | 0/5 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT05166603/Prot_SAP_000.pdf